CLINICAL TRIAL: NCT06605079
Title: Enhancing Palliative Care in ICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: European Commission (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and Intensive Care Medicine,Charité- University Berlin, Charite University, Berlin, Germany
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: EPIC
Record Dates: First submitted 2024-09-11; First posted 2024-09-20 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Palliative Care

STUDY DESIGN:
Intervention Model Description: Controlled, cluster-randomized, non-blinded, study in a stepped-wedge design with cross-over month.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intensive care unit patients in the intervention phase.
  Interventions: Behavioral: Complex intervention
- Control (Active Comparator): Intensive care unit patients with routine treatment in the control phase.
  Interventions: Other: Routine treatment

INTERVENTIONS:
Behavioral: Complex intervention — A complex intervention is carried out in the intensive care unit. This includes:
  * telemedical consultations by specialized palliative care experts from external institutions for the respective hospital staff
  * the training of hospital staff in the intensive care unit in basic palliative care and
  * the use of checklists for the early identification of eligible patients and the structured recording of palliative care needs.
  The efficacy and cost-effectiveness of the complex intervention will be investigated using a controlled clinical trial in a cluster-randomized controlled design. In addition, as part of the multicenter clinical study in WP 2 staff, patients and relatives will also be surveyed.
  Arms: Intervention
Other: Routine treatment — No complex intervention is established, just routine procedures.
  Arms: Control

SUMMARY:
The aim of this study is to reduce the suffering in intensive care through palliative care consultations.

DETAILED DESCRIPTION:
This project investigates the effectiveness and cost-effectiveness of palliative care consultations in the Intensive care unit. Charité will implement the Working Package 2 "Europe-wide harmonized and recommended palliative care practice for ICU" of the approved HORIZON funding application EPIC, to which this ethics application refers.

An accompanying anonymous employee survey (doctors/nurses) is conducted once in the intervention phase and once in the control phase in all study centers (see secondary endpoints 57-68 and 71).

ELIGIBILITY:
Patients:

Inclusion Criteria:

* Patients in ICU who can give consent and those who can not (via their authorized representative or legal guardian, also possible with delayed consent)
* From 18 years
* The leading cause of critical illness is not cancer
* New admission on the participating ICU > 72h
* Assessment of the need for palliative care by the in-charge physi-cian of the ICU, because (1) there is a significant disagreement about ICU treatment or (2) because the physician considers ther-apy limitations for the patient or (3) the physician considers a benefit from specialized PC consultation for ICU physician, nurse, or patient or family.

Exclusion Criteria:

- Patient is moribund and is expected to die within the next 24h

Study cohort relatives:

Inclusion criteria:

- At least one relative(s) of a patient. This may or may not be the legal representative, depending on national legislation.

Exclusion criteria:

* Refusal by the relative
* Refusal of the patient to participate in the intervention study
* <18 years of age

Cohort of employees:

Inclusion criteria

* Employed on the ITS as a doctor/nurse
* Employed in the clinical center as a member of the palliative care consultation service

Exclusion criterion Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2040 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Length of intensive care stay | During intensive care unit stay, an average of 5 days
  The primary endpoint is the number of days the patient spent in each Intensive Care Unit (ICU) of the index hospital during the first hospitalization.
  For example, if the patient was transferred from the first ICU participating in the EPIC study to another, second ICU within the same hospital, or if the patient was transferred back from a ward to the first ICU, the duration of the secondary ICU is included in the calculation of the primary endpoint.

SECONDARY OUTCOMES:
Costs | During intensive care unit stay, an average of 5 days
  Hospital cost and billing data, data on medical resource consumption combined with data on costs per unit of consumption at hospital level and from external sources, data on intervention costs including staff time for palliative care and related activities, hospital data or national data on salaries of individual professional groups.
Cost effectiveness | During intensive care unit stay, an average of 5 days
  Hospital data on salaries per occupational group
Readmissions to intensive care unit | During hospital stay, an expected average of 8 days
  The readmission rate of patients transferred out of the Intensive care unit
Maximum Sepsis-related organ failure assessment score (SOFA Score) in the intensive care unit | During intensive care unit stay, an average of 5 days
  To evaluate the performance of total maximum sequential organ failure assessment (SOFA) score and a derived measure, delta SOFA (total maximum SOFA score minus admission total SOFA) as a descriptor of multiple organ dysfunction/failure in intensive care.
Palliative Care assessment | During intensive care unit stay, an average of 5 days
  Presence of palliative care assessment performed during study period. The answer to the question: Has the palliative care assessment taken place? Yes/No
Presence of refractory symptoms I | During hospital stay, an expected average of 8 days
  Presence of refractory symptoms I is measured by physical symptoms.
Presence of refractory symptoms II | During intensive care unit stay, an average of 5 days
  Presence of refractory symptoms II is measured by distress of the patient.
Presence of refractory symptoms III | During intensive care unit stay, an average of 5 days
  Presence of refractory symptoms III is measured by distress of the family.
Presence of refractory symptoms IV | During intensive care unit stay, an average of 5 days
  Presence of refractory symptoms IV is measured by social problems of the patient.
Incidence of delirium | During intensive care unit stay, an average of 5 days
  Delirium is measured with validated delirium scores.
Presence and nature of treatment limitations | During intensive care unit stay, an average of 5 days
  Treatment limitation includes limits on the frequency of treatment, number of visits, days of coverage, or other similar limits on the scope or duration of treatment.
Length of hospital stay | During hospital stay, an average of 8 days
  Length of hospital stay is measured from ICU admission to discharge from hospital in days.
Informations on discharge | During hospital stay, an average of 8 days
  Where the patient is discharged to.
Informations on discharge | During intensive care unit stay, an average of 5 days
  Where the patient is discharged to.
Specialized palliative care expert | During hospital stay, an average of 8 days
  Presence of specialized palliative care expert consultation. Answer to the question: Was a specialized palliative care expert consulted? Yes/No Duration of measurement: Until hospital discharge
Mortality | Up to three months
  Intensive care unit, inhouse, until 30 days and until 3 months
Social Status of the patient | Up to three months
  The MacArthur Scale of Subjective Social Status (MacArthur SSS Scale) is a single-item measure that assesses a person's perceived rank relative to others in their group: To score this measure, researchers simply note the number of the rung (1-10) on which the respondent placed their "X."
Place of stay after hospitalization | Up to three months
  Place of stay after hospitalization is measured in questionnaire.
Home care after hospitalization | Up to three months
  Home care after hospitalization is measured in days.
Stress thermometer | Up to three months
  To measure psychological distress the German version of the National Comprehensive Cancer Network Distress Thermometer is used. The scale ranges from 0 (no distress) to 10 (extreme distress) with a cutoff score of 5, indicating a clinically significant level of distress.
Facilitators and barriers to high quality palliative care I | Up to three months
  Facilitators and barriers to high quality palliative care from the perspective of patients.
Facilitators and barriers to high quality palliative care II | Up to three months
  Facilitators and barriers to high quality palliative care from the perspective of relatives.
Symptom management by intensive care staff I | Up to three months
  Symptom management I by intensive care staff from the patient's perspective is measured with a questionnaire.
Symptom management by intensive care staff II | Up to three months
  Symptom management II by intensive care staff from the relative's perspective is measured with a questionnaire.
Treatment evaluation I | Up to three months
  Treatment evaluation I is measured from patients' perspective with a 5-point Likert scale (The choices range from Strongly Agree to Strongly Disagree).
Treatment evaluation II | Up to three months
  Treatment evaluation II is measured from the relatives' (proxy's) perspective with a 5-point Likert scale (The choices range from Strongly Agree to Strongly Disagree).
Evaluation of the provider's question about goals for treatment I | Up to three months
  Evaluation of the provider's question about goals for treatment I from the patients' perspective is measured with a 5-point Likert scale (The choices range from Strongly Agree to Strongly Disagree).
Evaluation of the provider's question about goals for treatment II | Up to three months
  Evaluation of the provider's question about goals for treatment II from the relatives' perspective is measured with a 5-point Likert scale (The choices range from Strongly Agree to Strongly Disagree).
Satisfaction with regard to communication I | Up to three months
  Satisfaction with regard to communication I from the patients' perspective is measured with a 5-point Likert scale (The choices range from Strongly Agree to Strongly Disagree).
Satisfaction with regard to communication II | Up to three months
  Satisfaction with regard to communication II from the relatives' perspective is measured with a 5-point Likert scale (The choices range from Strongly Agree to Strongly Disagree).
Evaluation of the quality of information regarding the treatment I | Up to three months
  Evaluation of the quality of information regarding the treatment from the patients' perspective is measured with a 5-point Likert scale (The choices range from Strongly Agree to Strongly Disagree).
Evaluation of the quality of information regarding the treatment II | Up to three months
  Rating of the quality of information regarding the treatment II from the relatives' perspective is measured with a 5-point Likert scale (The choices range from Strongly Agree to Strongly Disagree).
Suitability of care from the patient's perspective | Up to three months
  Suitability of care from the patient's perspective is measured with a 5-point Likert scale (The choices range from Strongly Agree to Strongly Disagree).
Outpatient resource utilization | Up to three months
  Outpatient resource utilization is measured by the number of outpatient visits.
Utilization of medical resources I | Up to three months
  Utilization of medical resources I is measured in days of mechanical ventilation.
Utilization of medical resources II | Up to three months
  Utilization of medical resources II is measured by Extracorporeal membrane oxygenation Yes/No.
Utilization of medical resources III | Up to three months
  Utilization of medical resources III is measured by dialysis Yes/No.
Utilization of medical resources IV | Up to three months
  Utilization of medical resources IV is measured by other organ replacement therapies. Yes/No.
Medical utilization after discharge from hospital I | During intensive care unit stay, an average of 5 days
  Medical utilization after discharge from hospital I is measured by number and days of re-hospitalizations in days.
Medical utilization after discharge from hospital II | Up to three months
  Medical utilization after discharge from hospital II is measured by days in care institutions in days.
Medical utilization after discharge from hospital III | Up to three months
  Medical utilization after discharge from hospital III is measured by outpatient healthcare encounters in days.
Medical utilization after discharge from hospital IV | Up to three months
  Medical utilization after discharge from hospital IV is measured by use of outpatient nursing services in days.
Medical utilization after discharge from hospital V | Up to three months
  Medical utilization after discharge from hospital V is measured by specialized outpatient palliative care (SAPV) in days.
Patient Health Questionnaire-4 I | Up to three months
  The Patient Health Questionnaire-4 (PHQ-4) I measures anxiety and depression in patients. The PHQ-4 is a four questionnaire answered on a four point Likert-type scale. A score of 3 or more on the depression/anxiety subscale is positive.
Patient Health Questionnaire-4 II | Up to three months
  The Patient Health Questionnaire-4 (PHQ-4) II measures anxiety and depression in relatives. The PHQ-4 is a four questionnaire answered on a four point Likert-type scale. A score of 3 or more on the depression/anxiety subscale is positive.
Health related quality of life I | Up to three months
  Health related quality of life I of the patient is measured with the 5-level EQ-5D version (EQ-5D-5L) from the EuroQol Group.
Question about the opinion of relatives on the unnecessary prolongation of life | Up to three months
  Question about the opinion of relatives on the unnecessary prolongation of life is measured by bipolar Likert scale.
Question about opinion of relatives on discomfort during the final hours before death | Up to three months
  Question about opinion of relatives on discomfort during the final hours before death is measured by bipolar Likert scale.
Question about opinion of relatives on loneliness during dying process. | Up to three months
  Question about opinion of relatives on loneliness during dying process is measured by bipolar Likert scale.
Patient and family friendliness of intensive care unit care I | Up to three months
  Patient and family friendliness of intensive care unit care I assessed by patients, measured with Likert scale/NRS 0-10).
Patient and family friendliness of intensive care unit care II | Up to three months
  Patient and family friendliness of intensive care unit care II assessed by relatives, measured by by Likert scale (too little, just right, too much)/NRS (0-10).
Informal care by relatives I | Up to three months
  Informal care by relatives I is measured by time spent with the patient.
Informal care by relatives II | Up to three months
  Informal care by relatives II is measured by impact on relative's income.
Informal care by relatives III | Up to three months
  Informal care by relatives III is measured by giving up relative´s professional activity.
Informal care by relatives IV | Up to three months
  Informal care by relatives IV is measured by reducing relative's professional activity.
Burnout Assessment Tool (BAT-12) | Up to 34 months.
  Twelve questions from the BAT-12 per employee based on 5 questions is measured with an electronic questionnaire once per intervention and once per control period.
Inappropriate therapy | Up to 34 months
  Perception of inappropriate therapy per employee based on 5 questions to employees is measured with an electronic questionnaire once per intervention and once per control period.
Moral distress | Up to 34 months
  Moral distress per employee is measured with numeric rating scale once per intervention and once per control period.
Implementation of the end-of-life practice | Up to 34 months
  Questions on the current implementation of the end-of-life practice based on 12 questions that are still being developed is measured with an electronic questionnaire once per intervention and once per control period.
Ethical decision-making climate in the intensive care unit | Up to 34 months
  Ethical decision-making climate in the intensive care unit per employee is measured with an electronic questionnaire once per intervention and once per control period.
Questions on the existence of Standard Operating Procedures | Up to 34 months
  Existence of Standard Operating Procedures per employee is measured with 4 questions with an electronic questionnaire once per intervention and once per control period.
Questions about using the ABCDEF bundle | Up to 34 months
  Questions about using the ABCDEF bundle is measured with 11 questions with an electronic questionnaire once per intervention and once per control period.
Questions about supporting measures | Up to 34 months
  Questions about supporting measures is measured with 4 questions with an electronic questionnaire once per intervention and once per control period.
Perception of palliative care and law | Up to 34 months
  Perception of palliative care and law is measured with 4 questions with an electronic questionnaire once per intervention and once per control period.
Question about hurdles to palliative care | Up to 34 months
  Question about hurdles to palliative care in the intensive care medicine is measured with 1 question with an electronic questionnaire once per intervention and once per control period.
Question about supporting factors | Up to 34 months
  Question about supporting factors to palliative care in the intensive care medicine is measured with 1 question with an electronic questionnaire once per intervention and once per control period.
Comments after beginning of the intervention phase | Up to 34 months
  Comments can be made via free text in an electronic questionnaire once per intervention and once per control period.

OTHER OUTCOMES:
Demographic data of the patients | During intensive care unit stay, an average of 5 days
  Demographic data of the patient (age, gender, main diagnosis and reasons for intensive care, insurance status, religion yes/no, highest level of education, employment status, existence of living will, patient power of attorney, chronic conditions) are measured with a questionnaire.
Demographic data of the relatives | Up to three months
  Demographic data of the relative (age, gender, relationship to the patient, representative/guardian, religion yes/no) are measured with a questionnaire.
Employee demographics | Up to 34 months
  Employee demographics (age group, gender, profession, years of professional experience, years and experience in palliative care and/or ethical training, type of intensive care unit) are measured with an electronic questionnaire once per intervention and once per control period.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charité-University Medicine (Berlin, Germany); Martin Neukirchen, MD, Study Director — Heinrich-Heine-University Düsseldorf, Germany; Jochen Dutzmann, MD, Study Director — University Medicine Halle, Germany; Spyros Mentzelopoulos, MD, Prof., Study Director — National and Kapodistrian University of Athens, Greece; Katerina Rusinova, MD, Study Director — Charles University in Prague, Italy; Akiva Nachshon, MD, Study Director — Hebrew University of Jerusalem, Israel; Edoardo de Robertis, MD, Prof., Study Director — University Of Perugia
Locations (31):
- Czechia (3):
  - ICU General Resuscitation (RES UP), General University hospital, Prague
  - ICU General Resuscitation (RES2), Prague
  - ICU Metabolic, General University hospital, Prague
- Germany (13):
  - Department of Anesthesiology and Intensive Care Medicine (CCM/CVK),Charité - University Medicine Berlin, Mitte, State of Berlin
  - Department of Anesthesiology and Intensive Care Medicine (CCM/CVK),Charité - University Medicine Berlin, Wedding, State of Berlin
  - CARITAS Klinik Maria Heimsuchung, Berlin
  - Charité - Department of Anesthesiology and Intensive Care Medicine CBF, Berlin
  - Department of Cardiology, Angiology and Intensive Care Medicine | CVK, Charité - University Berlin, Berlin
  - Evangelisches Krankenhaus Hubertus, Berlin
  - Unfallkrankenhaus Berlin, Berlin
  - Medical and Neurological Intensive Care Unit, University Hospital of Düsseldorf, Düsseldorf
  - Neurosurgical and Traumatological ICU ZI13, University Hospital of Düsseldorf, Düsseldorf
  - Surgical Intensive Care Unit CIA1/CIB1, University Hospital of Düsseldorf, Düsseldorf
  - Universitätsklinikum Halle (Saale): Klinik für Innere Medizin III, Halle
  - Johanna-Etienne Hospital Neuss, Interdisciplinary ICU, Neuss
  - Ev. Krankenhaus Paul-Gerhardt-Stift Wittenberg:Angiologie und Kardiologie, Wittenberg
- Greece (8):
  - Department of Intensive Care Medicine, University Hospital of Heraklion, Heraklion, Crete
  - Department of Intensive Care Medicine, University Hospital of Patras, Pátrai, Rio
  - Department of Intensive Care Medicine, University Hospital of Alexandroupolis, Alexandroupoli
  - Cardiothoracic Intensive Care Unit of the Onassis Cardiac Surgery Center, Athens
  - Department of Intensive Care Medicine, Alexandra General Hospital, Athens
  - Department of Intensive Care Medicine, Evaggelismos General Hospital, Athens
  - Department of Intensive Care Medicine, University Hospital of Ioannina, Ioannina
  - University Hospital of Larissa, Critical Care Department, Larissa
- Israel (3):
  - General Intensive Care Unit, Hadassah Medical Organisation, Jerusalem
  - The Coronary Care Intensive Care Unit, Hadassah Hospital, Ein Kerem, Jerusalem
  - The Neurosurgical Intensive Care Unit, Hadassah Hospital, Ein Kerem, Jerusalem
- Italy (4):
  - S.C. Anestesia e Rianimazione 1 - Terapia Intensiva Cardiochirurgica, Azienda Ospedaliera Universitaria S. Maria della Misericordia, Perugia
  - S.C. Anestesia e Rianimazione 2 - Terapia Intensiva, Azienda Ospedaliera Universitaria S. Maria della Misericordia, Perugia
  - UOC di Anestesia e Rianimazione Cardio Toraco Vascolare dell'AOU San Giovanni di Dio e Ruggi d'Aragona "Scuola Medica Salernitana", Salerno University Hospital, Salerno
  - S.C. Anestesia - Rianimazione Azienda Ospedaliera Santa Maria - Terni, Terni

IPD SHARING:
Plan to Share IPD: No